CLINICAL TRIAL: NCT05805891
Title: An Exploratory Clinical Study on Bortezomib for the Treatment of Refractory Rheumatoid Arthritis
Brief Title: Bortezomib for the Treatment of Refractory Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese SLE Treatment And Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bortezomib-RA
Record Dates: First submitted 2023-03-22; First posted 2023-04-10 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-03

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; bortezomib
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Bortezomib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bortezomib (Experimental): bortezomib added on previous treatment
  Interventions: Drug: bortezomib

INTERVENTIONS:
Drug: bortezomib — bortezomib 2mg/week subcutaneous injection

SUMMARY:
This is a single-center, single-arm, prospective study on the efficacy and safety of Bortezomib in addition to standard therapy in patients with refractory rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18~70 years.
2. Fulfilling the 2010 ACR/EULAR classification criteria for RA.
3. Failed to at least two bDMARDs (including but not limited to TNF inhibitors, IL-6 receptor inhibitors, T cell costimulation inhibitor and anti-B cell biologics) or tsDMARDs (including but not limited to JAK inhibitors) in combination with a csDMARD for at least 12 weeks. The dosage of cs/b/tsDMARDs needs to be stable for at least 6 weeks.
4. For patients receiving glucocorticoids, the dosage of GC needs to be less than or equal to 10mg prednisone equivalent and stable for at least 6 weeks.
5. For patients receiving non-steroid anti-inflammatory drugs, the dosage of NSAID needs to be stable for at least 2 weeks.
6. Neutrophil≥1.0×10^9/L, platelet≥100×10^9/L, alanine transaminase (ALT) and aspartate aminotransferase (AST) within 3 ULN, total bilirubin within 1.5 ULN.
7. Informed consent obtained.

Exclusion Criteria:

1. Other concomitant autoimmune diseases (except for Sjogren's syndrome secondary to rheumatoid arthritis).
2. The presence of severe uncontrolled cardiovascular, cerebrovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological or neuropsychiatric disorders, or abnormal laboratory tests. The investigators consider that participation in the study may make unacceptable risks to the subjects.
3. A history of malignancy with a clinical cure time of less than 5 years.
4. Pregnant or breast-feeding women, or planning to get pregnant or start breastfeeding during the study.
5. Vaccinated with live attenuated virus within 4 weeks before entering the study.
6. Allergic to bortezomib or mannitol.
7. Participated in any other investigational drug trial within 12 weeks before study initiation.
8. Active hepatitis or liver disease at the time of screening: Hepatitis B surface antigen (HBsAg) or anti-hepatitis C virus antibodies (HCVAb) positive; (Note: If Hepatitis B Core Antibody, (HBcAb) is positive and HBsAg is negative, HBV-DNA detection will be performed, patient is eligible if HBV-DNA was negative).
9. Active herpes zoster infection, or severe infection requiring intravenous antibiotics or hospitalization occurred 12 weeks before study initiation.
10. Other conditions that not suitable for inclusion in the study, assessed by the investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
DAS28 remission or LDA at week 24 | 24 weeks
  Proportion of patients who achieve remission or low disease activity (LDA) at week 24 according to DAS 28.

SECONDARY OUTCOMES:
DAS28 improvement at week 12 | 12 weeks
  Proportion of patients who achieve remission or low disease activity at week 12 according to DAS 28. Proportion of patients who achieve at least a 50% reduction of DAS28 at week 12.
SDAI improvement at week 12 and remission or LDA at week 24 | 24 weeks
  Proportions of patients who achieve remission or low disease activity at week 12 and week 24 according to SDAI. Proportion of patients who achieve at least a 50% reduction of SDAI at week 12.
CDAI improvement at week 12 and remission or LDA at week 24 | 24 weeks
  Proportions of patients who achieve remission or low disease activity at week 12 and week 24 according to CDAI. Proportion of patients who achieve at least a 50% reduction of CDAI at week 12.
ACR20, ACR50 and ACR70 at week 12 and week 24 | 24 weeks
  Proportions of patients who achieve ACR20, ACR50 and ACR70 at week 12 and week 24.
Changes in glucocorticoid dose | 24 weeks
  Changes in glucocorticoid dose at week 12 and 24 from baseline.
Adverse events during the study | 28 weeks
  All adverse events, severe adverse events and proportion of patients who discontinued bortezomib due to adverse events from the first dose of bortezomib to 4 weeks after the last dose.

CONTACTS AND LOCATIONS:
Overall Officials: Xinping Tian, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided